CLINICAL TRIAL: NCT02199847
Title: An Evaluation of the Effects of Pharmaton® Caplets Film-coated Tablets on Mental Performance and Physical Fatigue in Nurses Working Night Shifts: a Double-blind, Placebo Controlled Pilot Trial
Brief Title: Evaluation of the Effects of Pharmaton Tablets on Mental Performance and Physical Fatigue in Nurses Working Night Shift
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1114.11
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Sleep Disorders, Circadian Rhythm
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

ARMS (2):
- Pharmaton® Caplets (Experimental)
  Interventions: Drug: Pharmaton® Caplets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pharmaton® Caplets
  Arms: Pharmaton® Caplets
Drug: Placebo
  Arms: Placebo

SUMMARY:
The general aim of this study is to assess the effects of Pharmaton® Caplets on mental performance and physical fatigue in nurses and nursing auxiliaries working night shifts

ELIGIBILITY:
Inclusion Criteria:

* Male and female nurses and nursing auxiliaries working night shift
* Age range: 20 to 45 inclusive
* BMI range: 18-30
* Negative pregnancy test for females
* Subjects must be free of any clinically significant disease or condition that required a physician's care and/or was to interfere with study evaluation and procedures
* Clinical laboratory tests within normal limits or, if out of normal range, clinically acceptable to the investigator
* Negative urine drug screen for drugs at screening
* Subjects must be willing to give informed consent prior to study enrolment and be able to adhere to restrictions and examination schedules

Exclusion Criteria:

* Any serious disorder that may interfere with his/her participation to the trial and the evaluation of the safety of the test drug (e.g. liver and/or renal disease, hypervitaminosis A, psychic disorder, etc.) and/or treatment with chronic medication
* Pre-treatment (less than 2 weeks prior to inclusion in this trial) and/or concomitant treatment with any drug that may influence the trial symptomatology and may interfere with evaluation of the safety of the test drug (e.g. vitamins and minerals supplementation)
* Individuals drinking more than 40 g alcohol/day (glass of 12.5 cl of wine 10° = 12 g; glass of 4 cl of aperitif 42° = 17 g; glass of 25 cl of beer 3° = 7.5 g; glass of 25 cl of beer 6° = 15 g); Alcohol and drug abuse according to Diagnostic and Statistic Manual, Version IV (DSM-IV)
* Individuals drinking more that 6 cups of coffee or tea/day
* Individuals smoking more than 10 cigarettes/day
* Female volunteers in child-bearing age not using adequate means of birth control (contraceptive pills, Intrauterine Device (IUD), sterilization)
* Pregnancy and/or lactation
* Relevant allergy or known hypersensitivity to the investigational product or its excipients
* Individuals taking or having taken recently other vitamins and minerals supplementation
* Individuals with a current disorder likely to modify EEG recordings and/or computerized cognitive testing
* Individuals having a history of cancer
* Participation in another clinical trial within the last 3 months prior to the start of the study and concurrent participation in another clinical trial
* Individuals without health insurance

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2000-06; Primary Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mental performance as measured by the completion of Cognitive Drug Research tasks (CDR tasks) combined with Electroencephalogram (EEG) (post-shift) | at day 77

SECONDARY OUTCOMES:
Change in mental performance as measured by the completion of Cognitive Drug Research tasks (CDR tasks) combined with Electroencephalogram) | up to day 77
Assessment of spontaneous Electroencephalogram (EEG) and event related potentials | up to day 77
Assessment of Sleep-Electroencephalogram parameters | Day -1, Day 1, Day 77
Evaluation of Quality of life scales | up to day 77
Evaluation of Sleep by Visual Analogue Scale (VAS) | up to day 77
Assessment of 24-hours holter Electrocardiogram (ECG) | Day -1, Day1, Day 77
Assessment of urinary cortisol levels | Day -1, Day1, Day 77
Number of patients with adverse events | up to 3 months
Assessment of tolerability by investigator on a 4-point scale | at day 77
Assessment of tolerability by subject on a 4-point scale | Day 41, Day 77